CLINICAL TRIAL: NCT00393432
Title: Enhancing Motor Memory Encoding by Action Observation
Brief Title: Enhancing Motor Task Training by Action Observation Watching Others Perform the Task
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070010; 07-N-0010
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-18

CONDITIONS: Motor Memory
Keywords: Action Observation; Motor Memory; Transcranial Magnetic Stimulation (TMS); Use-Dependent Plasticity; Healthy Volunteer; HV

SUMMARY:
This study will determine how the brain learns a new motor task when the subject practices the task and watches others perform it (action observation) at the same time.

Healthy normal volunteers between 18 and 55 years of age may be eligible for this study. Candidates are screened with a medical history, general and neurological exam, and a brain MRI if one has not been done within 12 months of entering the study. Participants undergo one or both of the following experiments:

1. Effect of Transcranial Magnetic Stimulation on Motor Training and Action Observation

   Subjects participate in at least 12 4-hour test sessions, separated by at least 1 day. Each session includes the following:
   * Functional MRI (fMRI): MRI scanning uses a magnetic field and radio waves to produce images of the brain. For fMRI, the subject performs tasks during the scan to allow researchers to see brain changes that occur during performance of the activity.
   * Transcranial magnetic stimulation (TMS): For this test, a wire coil is held on the scalp. A brief electrical current passes through the coil to stimulate the brain. The stimulation may cause a twitch in muscles of the face, arm, or leg, and the subject may hear a click and feel a pulling sensation on the skin under the coil. During the stimulation, the subject is asked to: 1) perform the training task (make brisk thumb movements); 2) watch a video showing the hand of another person performing the same task; and 3) perform the task and watch the video at the same time, synchronizing his or her movements with those observed in the video.
   * Surface electromyography: Electrodes are filled with a conductive gel and taped to the skin over a hand muscle to measure the electrical activity of the muscle.
   * Behavioral measurements: Evaluation of learned movement tasks.
   * Questionnaires to test attention, fatigue and mood before, during and after each test session.
2. Effect of Pharmacological Agents on Motor Training and Action Observation

Subjects participate in no more than 12 5-hour test sessions, separated by at least 2 days. In the course of the 12 sessions, subjects receive each of three medications - dextromethorphan, scopolamine and rivastigmine - three times and a placebo (pill with no active ingredient) three times. During each session, subjects have TMS measurements, behavioral measurements and electromyography as described in experiment 1.

DETAILED DESCRIPTION:
Motor training (MT) elicits formation of motor memories in the human primary motor cortex. Observing another individual perform motor training (Action Observation, AO) also results in formation of motor memories in M1. AO enhances motor training effects (MT+AO) on the formation of motor memories. Possible underlying mechanisms include long-term potentiation (LTP), a process influenced by N-methyl-D-aspartate (NMDA) receptor activation, gamma-aminobutyric acid (GABA), norepinephrine (NE), dopamine and acetylcholine (Ach), taking place at the confluence of inputs from PMv over the primary motor cortex (M1).

The purpose of this protocol is to gain insight into the mechanisms underlying motor memory formation by MT+AO. We plan to perform two different types of experiments: In experiment 1, we will modulate activity in PMv using TMS to investigate the role of this cortical area on motor memory formation induced by MT+AO. In experiment 2, we will test the effects of single doses of (a) the NMDA receptor antagonist dextromethorphan, (b) the muscarinic receptor antagonist scopolamine, both known to disrupt LTP, and (c) the cholinesterase inhibitor rivastigmine, which enhances LTP.

The primary outcome measure of motor memory formation will be the percentage of TMS-evoked movements that fall within the training target zone (TTZ) before and after MT+AO. The secondary outcome measure will be the percentage of TMS-evoked movements that fall within TTZ before and after MT alone and AO alone.

Expected results are (1) upregulation of activity in PMv using 0.1 Hz TMS will enhance motor memory formation induced by MT+AO more than sham TMS and downregulation of PMv using 0.9 Hz TMS and (2) dextromethorphan and scopolamine will decrease but rivastigmine will increase motor memory formation induced by MT+AO with placebo. This study may provide useful information on the mechanisms underlying the beneficial effects of action observation on neuroplasticity.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age between 18-55 years
  2. Able to perform tasks required by the study
  3. Willing and able to give consent
  4. Possibility to obtain TMS-evoked thumb movements in a consistent direction at baseline

EXCLUSION CRITERIA:

Subjects are not eligible for this experiment if they:

1. Are unable to perform the tasks
2. Have history of severe alcohol or drug abuse, psychiatric illness like severe depression and poor motivational capacity
3. Have problems with movement of the hands
4. Are receiving drugs acting primarily on the central nervous system
5. Are pregnant
6. Have medical or technical contraindications to MRI procedures or devices producing artifacts that impair MRI signal (e.g., dental braces, pacemakers, implanted medication pumps, cochlear devices, neural stimulators, metal in the cranium, surgical clips, and other metal/magnetic implants, claustrophobia)
7. Have had an allergic reaction to scopolamine. Have glaucoma, severe liver disease, kidney disease, an enlarged prostrate gland or a blocked digestive tube
8. Have had an allergic reaction to dextromethorphan
9. Are using a MAO inhibitor (such as Parnate [registered trademark], Nardil [registered trademark], or Marplan [registered trademark] or if you have used one of these drugs in the past 2 weeks
10. Have asthma
11. Are taking pain or arthritis medicine (sometimes called NSAIDs) such as aspirin, ibuprofen, or naproxen on a regular basis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2006-10-18; Study Completion 2008-07-18

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Apland JP, Braitman DJ. Effects of non-opioid antitussives on epileptiform activity and NMDA responses in hippocampal and olfactory cortex slices. Brain Res. 1990 Oct 8;529(1-2):277-85. doi: 10.1016/0006-8993(90)90838-3. PMID 2282497
- [Background] Buccino G, Binkofski F, Fink GR, Fadiga L, Fogassi L, Gallese V, Seitz RJ, Zilles K, Rizzolatti G, Freund HJ. Action observation activates premotor and parietal areas in a somatotopic manner: an fMRI study. Eur J Neurosci. 2001 Jan;13(2):400-4. PMID 11168545
- [Background] Butefisch CM, Khurana V, Kopylev L, Cohen LG. Enhancing encoding of a motor memory in the primary motor cortex by cortical stimulation. J Neurophysiol. 2004 May;91(5):2110-6. doi: 10.1152/jn.01038.2003. Epub 2004 Jan 7. PMID 14711974